CLINICAL TRIAL: NCT06078202
Title: Assessment of the Relative Bioavailability of Three Immediate-Release Tablet Formulations of ABBV-903 in Healthy Volunteers
Brief Title: A Study to Assess the Relative Bioavailability of Three Immediate-Release Tablet Formulations of ABBV-903 in Healthy Adult Volunteers
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Strategic considerations
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M24-231
Record Dates: First submitted 2023-10-05; First posted 2023-10-11 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Healthy Volunteers
Keywords: ABBV-903; Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Part 1, Sequence A (Experimental): Participants will receive 1 dose of ABBV-903.
  Interventions: Drug: ABBV-903
- Part 1, Sequence B (Experimental): Participants will receive 1 dose of ABBV-903.
  Interventions: Drug: ABBV-903
- Part 1, Sequence C (Experimental): Participants will receive 1 dose of ABBV-903.
  Interventions: Drug: ABBV-903
- Part 2, Sequence A (Experimental): Participants will receive 1 dose of ABBV-903.
  Interventions: Drug: ABBV-903
- Part 2, Sequence B (Experimental): Participants will receive 1 dose of ABBV-903.
  Interventions: Drug: ABBV-903

INTERVENTIONS:
Drug: ABBV-903 — Tablet; oral

SUMMARY:
The purpose of this study is to evaluate the relative bioavailability of three immediate-release table formulations of ABBV-903 under fasting conditions in healthy volunteers, and to evaluate the effect of food on the pharmacokinetics of three immediate-release table formulations of ABBV-903.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) is >= 18.0 to <= 32.0 kg/m2 after rounding to the tenths decimal, at screening and upon initial confinement.
* A condition of general good health, based upon the results of a medical history, physical examination, vital signs, laboratory profile and a 12-lead electrocardiogram (ECG).

Exclusion Criteria:

* History of any clinically significant illness/infection/major febrile illness, hospitalization, or any surgical procedure within 30 days prior to the first dose of study drug.
* History of epilepsy, any clinically significant cardiac, respiratory (except mild asthma as a child), endocrine, renal, hepatic, gastrointestinal, hematologic or psychiatric disease or disorder, or any uncontrolled medical illness.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of ABBV-903 | From 0 - 96 hours
  Cmax of ABBV-903 will be assessed.
Time to Cmax (Tmax) of ABBV-903 | From 0 - 96 hours
  Tmax of ABBV-903 will be assessed.
Apparent Terminal Phase Elimination Constant (BETA) of ABBV-903 | From 0 - 96 hours
  BETA of ABBV-903 will be assessed.
Terminal Phase Elimination Half-life (t1/2) of ABBV-903 | From 0 - 96 hours
  Terminal phase elimination half-life (t1/2) of ABBV-903 will be assessed.
Area Under the Plasma Concentration-time Curve from Time 0 until 24 Hours after Dosing (AUC0-24) of ABBV-903 | From 0 - 96 hours
  AUC0-24 of ABBV-903 will be assessed.
AUC from Time 0 until the Last Measurable Concentration (AUCt) of ABBV-903 | From 0 - 96 hours
  AUCt of ABBV-903 will be assessed.
AUC from Time 0 to Infinite Time (AUCinf) of ABBV-903 | From 0 - 96 hours
  AUCinf of ABBV-903 will be assessed.
Number of Participants with Adverse Events | Up to 42 days
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (1):
- Acpru /Id# 259438, Grayslake, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M24-231